CLINICAL TRIAL: NCT04967638
Title: Survival Analysis of Segmental Mandibulectomy With Immediate Vascularized Fibula Flap Reconstruction in Stage IV Oral Squamous Cell Carcinoma Patients
Brief Title: Survival Analysis of Oral Cancer Patients
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Hongyang Ma, Doctor, KU Leuven
Other Study IDs: S63615-1
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Head and Neck Cancer
Keywords: Squamous cell carcinoma; Free fibula flap; Prognosis; Survival; Mandibular reconstruction
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: tumor resection and mandible reconstruction — The patients who underwent primary ablative tumor resection with segmental mandibulectomy and immediate VFF reconstruction were retrieved from the database

SUMMARY:
This study aims to assess the survival rate of oral squamous cell carcinoma (OSCC) patients following immediate mandibular reconstruction with vascularized fibula flap (VFF) and to identify risk factors influencing the overall survival rate and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stage IV OSCC
* Follow-up period more than one year.

Exclusion Criteria:

* Non-neoplastic diseases
* Two-staged reconstruction
* Presurgical distant metastasis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The files of patients diagnosed and treated between January 1996 to June 2019 for OSCC were retrospectively reviewed. The patients who underwent primary ablative tumor resection with segmental mandibulectomy and immediate VFF reconstruction were retrieved from the database
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
The overall cumulative survival | 5th year
  The overall cumulative survival was recorded at the fifth-year.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No